CLINICAL TRIAL: NCT03443115
Title: Multicenter Cohort Study on Duchenne Muscular Dystrophy Cardiomyopathy
Brief Title: Duchenne Muscular Dystrophy Heart Study
Acronym: DMD-HS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hôpital Cochin (Other)
Collaborators: Association Monégasque contre les Myopathies (Unknown)
Responsible Party: Principal Investigator, Karim Wahbi, MD, PhD, Hôpital Cochin
Other Study IDs: DMD-HS
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Duchenne Muscular Dystrophy; Duchenne Muscular Dystrophy-Associated Dilated Cardiomyopathy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective cohort study including patients with genetically proven Duchenne muscular dystrophy, diagnosed from January 1993 to March 2020.

Inclusion of the data relative to genetic diagnosis, clinical characteristics at baseline, cardiac and respiratory workup, medical treatments (ACE inhibitors, steroids), surgical procedures, and occurrence during follow-up of cardiac, respiratory and fatal events.

Objectives are to describe long-term natural history of the disease, vital prognosis, genotype-phenotype correlations, effect of treatments.

ELIGIBILITY:
Inclusion Criteria:

* Genetically-proven Duchenne Muscular Dystrophy (DMD mutation)
* Covering by social security

Exclusion Criteria:

* Patient refusal to participate to the study

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients diagnosed with Duchenne muscular dystrophy and referred to reference centers for neuromuscular diseases for the management of their condiction.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2017-06-27 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | Follow-up completed in March 2020

SECONDARY OUTCOMES:
Hospitalization for heart failure | Follow-up completed in March 2020
Dilated cardiomyopathy | Follow-up completed in March 2020
Hospitalization for acute respiratory failure | Follow-up completed in March 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Cochin Reference Center for Neuromuscular Diseases, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Porcher R, Desguerre I, Amthor H, Chabrol B, Audic F, Rivier F, Isapof A, Tiffreau V, Campana-Salort E, Leturcq F, Tuffery-Giraud S, Ben Yaou R, Annane D, Amedro P, Barnerias C, Becane HM, Behin A, Bonnet D, Bassez G, Cossee M, de La Villeon G, Delcourte C, Fayssoil A, Fontaine B, Godart F, Guillaumont S, Jaillette E, Laforet P, Leonard-Louis S, Lofaso F, Mayer M, Morales RJ, Meune C, Orlikowski D, Ovaert C, Prigent H, Saadi M, Sochala M, Tard C, Vaksmann G, Walther-Louvier U, Eymard B, Stojkovic T, Ravaud P, Duboc D, Wahbi K. Association between prophylactic angiotensin-converting enzyme inhibitors and overall survival in Duchenne muscular dystrophy-analysis of registry data. Eur Heart J. 2021 May 21;42(20):1976-1984. doi: 10.1093/eurheartj/ehab054. PMID 33748842